CLINICAL TRIAL: NCT02037919
Title: Immediate vs. Delayed Insertion of Nexplanon After Termination of Pregnancy Over 14-weeks Gestation (NAPA)
Brief Title: Nexplanon Application Post-Abortion (NAPA)
Acronym: NAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Family Planning Associates Medical Group, LTD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Allison Cowett, MD MPH, Associate Medical Director, Family Planning Associates Medical Group, LTD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIS#50302: Women's Health MISP
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Contraception; Abortion, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Nexplanon Insertion (Experimental): An etonogestrel rod will be placed within 15 minutes following the abortion procedure.
  Interventions: Other: Immediate Nexplanon Insertion
- Post-op Nexplanon Insertion (Active Comparator): Participants in the "delayed" placement group will be asked to return to Magee-Womens Hospital for a post-abortion visit 2-4 weeks following the procedure. Participants in the delayed group will be offered a method of contraception to use in the interim between their procedure and their insertion appointment. At this time an etonogestrel rod will be placed in her arm using standard procedure.
  Interventions: Other: Post-op Nexplanon Insertion

INTERVENTIONS:
Other: Immediate Nexplanon Insertion — Patient will have a Nexplanon inserted within 15 minutes of her abortion
  Arms: Immediate Nexplanon Insertion
Other: Post-op Nexplanon Insertion — Place Nexplanon at post operative visit rather than at surgery
  Arms: Post-op Nexplanon Insertion

SUMMARY:
Women who receive Nexplanon immediately post abortion will be significantly more likely to be using the device 6 months after the procedure than those assigned to receive the device 2-4 weeks after the procedure.

DETAILED DESCRIPTION:
Women will be contacted 6 months after their abortion to ask about contraception use and side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older,
* an intrauterine pregnancy > 14 weeks and <23 6/7 weeks gestation and desire termination of pregnancy
* desire a Nexplanon for contraception
* able to give informed consent in English
* no contraindications to Nexplanon (based on U.S. CDC Medical Eligibility Criteria for Contraception) or D&E

Exclusion Criteria:

* unable to give informed consent
* have any of the following medical conditions: active venous thromboembolism, known or suspected sex-steroid sensitive malignancies, current hepatic disease with abnormal liver function tests, undiagnosed vaginal bleeding, hypersensitivity to any of the ingredients in Nexplanon.
* non-surgical management of pregnancy
* prior participation in this study
* breast cancer or a history of breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Cremer, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Family Planning Associates Medical Grooup, LTD, Chicago, Illinois
  - University of Pittsburgh, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 148 participants were recruited and randomized into two study arms.
Pre-assignment Details: Participants were randomized.
Period: Overall Study
Arm/Group | Immediate Nexplanon Insertion | Post-op Nexplanon Insertion
Started | 73 (Randomized to immediate insertion) | 75 (32 participants had implants inserted)
Had Implant Inserted | 73 | 32
Contacted at Six Months and Using Implant | 40 | 19
Contacted at 6 Months and Not Using Implant | 3 (Had implant removed) | 11 (3 participants had implant removed 8 participants never had implant inserted)
Completed (Contacted at 6 months and completed telephone follow up) | 43 | 30
Not Completed | 30 | 45
Not completed — Lost to Follow-up | 30 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Nexplanon Insertion | Post-op Nexplanon Insertion | Total
Number analyzed (Participants) | 73 | 75 | 148
Age, Continuous [Median (Full Range); unit: years] | 25 [18 to 41] | 23 [18 to 40] | 24 [18 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 75 | 148
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 28 | 22 | 50
  Race: African American | 45 | 52 | 97
  Race: Native American or Alaska Native | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73 | 75 | 148
Education [Count of Participants; unit: Participants]
  Less than high school | 10 | 14 | 24
  High school equivalency certificate | 27 | 25 | 52
  Some college | 28 | 31 | 59
  Associate's degree | 5 | 2 | 7
  Bachelor's degree | 3 | 3 | 6
Marital Status [Count of Participants; unit: Participants]
  Never married | 69 | 70 | 139
  Married | 2 | 2 | 4
  Separated or divorced | 2 | 3 | 5
Positive Smoking Status [Count of Participants; unit: Participants] | 17 | 15 | 32
Insurance Type [Count of Participants; unit: Participants]
  None | 20 | 10 | 30
  Public | 50 | 57 | 107
  Private | 3 | 7 | 10
  Private and Public | 0 | 1 | 1
Using insurance for D&E [Count of Participants; unit: Participants]
  Yes | 1 | 3 | 4
  No | 20 | 11 | 31
  Not Covered | 52 | 61 | 113
Latina [Count of Participants; unit: Participants] | 22 | 20 | 42
Total no. of pregnancies [Median (Full Range); unit: Number of pregnancies]
  Total | 4 [1 to 12] | 4 [1 to 10] | 4 [1 to 12]
  Term | 1 [0 to 8] | 1 [0 to 8] | 1 [0 to 8]
  Preterm | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 2]
  Abortion | 1 [0 to 5] | 1 [0 to 4] | 1 [0 to 5]
No. of children alive [Median (Full Range); unit: Number of children alive] | 2 [0 to 8] | 1 [0 to 8] | 1.5 [0 to 8]
Prior D&E [Count of Participants; unit: Participants] | 36 | 41 | 77
D&E indication [Count of Participants; unit: Participants]
  Social or economic | 59 | 61 | 120
  Fetal anomaly | 0 | 2 | 2
  Maternal health issue | 2 | 4 | 6
  Other | 15 | 15 | 30
  Declined to answer | 2 | 2 | 4
Birth control methods used in the past [Count of Participants; unit: Participants]
  Implant | 3 | 3 | 6
  LNG IUD | 5 | 5 | 10
  Pill, patch, or ring | 55 | 52 | 107
  DMPA | 42 | 45 | 87
  Barrier | 71 | 71 | 142
  Abstinence | 4 | 1 | 5
  Withdrawal | 14 | 21 | 35
  None | 1 | 3 | 4
History of STI [Count of Participants; unit: Participants] | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Intention-to-treat Analysis of Etonogestrel Implant Use
Description: Current use of Etonogestrel implant, confirmed via phone by participant palpation, at 6 months post-insertion, with all entire sample used in calculations.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Nexplanon Insertion | Post-op Nexplanon Insertion
Number analyzed (Participants) | 73 | 75
Participants
  Using implant at 6 months | 40 | 19
  Implant removed before 6 months | 3 | 3

2. Primary Outcome: Per-protocol Analysis of Etonogestrel Implant Use
Description: Current use of Etonogestrel implant, confirmed via phone by participant palpation, at 6 months post-insertion, with only participants who completed the 6-month follow-up used in calculations.
Time Frame: 6 months
Population: Calculated using only participants who completed the 6-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Nexplanon Insertion | Post-op Nexplanon Insertion
Number analyzed (Participants) | 43 | 30
Participants
  Using implant at 6 months | 40 | 19
  Implant removed before 6 months | 3 | 3
  Implant never placed | 0 | 8

3. Secondary Outcome: Repeat Pregnancy
Description: Occurrence of a pregnancy within 6 months after second-trimester abortion.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Nexplanon Insertion | Post-op Nexplanon Insertion
Number analyzed (Participants) | 43 | 30
Participants
  Repeat pregnancy within 6 months | 1 | 1
  No repeat pregnancy in 6 months | 42 | 29

4. Other Pre Specified Outcome: Implant Inserted
Description: Whether participants had the implant inserted as part of the study
Time Frame: Within 4 weeks of abortion
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Nexplanon Insertion | Post-op Nexplanon Insertion
Number analyzed (Participants) | 73 | 75
Participants | 73 | 32

5. Other Pre Specified Outcome: Completed 6-month Phone Call
Description: Whether participants completed 6-month phone call follow-up.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Nexplanon Insertion | Post-op Nexplanon Insertion
Number analyzed (Participants) | 73 | 75
Participants | 43 | 30

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Post-op Nexplanon Insertion: Participants in the "delayed" placement group will be asked to return to Family Planning Associates for a post-abortion visit 2-4 weeks following the procedure. Participants in the delayed group will be offered a method of contraception to use in the interim between their procedure and their insertion appointment. At this time an etonogestrel rod will be placed in her arm using standard procedure.
  Post-op Nexplanon Insertion: Place Nexplanon at post operative visit rather than at surgery
Arm/Group | Immediate Nexplanon Insertion | Post-op Nexplanon Insertion
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/75
Other Adverse Events (participants affected / at risk) | 2/73 | 1/75
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Nexplanon Insertion (N=73) | Post-op Nexplanon Insertion (N=75)
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3)
Rapid weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Post abortal endometritis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pregnancy (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-01-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT02037919/Prot_SAP_000.pdf
  • Informed Consent Form (2015-10-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT02037919/ICF_001.pdf